CLINICAL TRIAL: NCT06466928
Title: A Nationwide Analysis of Total Pancreatectomy
Brief Title: Total Pancreatectomies in Germany - Epidemiology, Trends,
Acronym: ToPaGe
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: Margarete-Ammon-Stiftung (Unknown)
Responsible Party: Principal Investigator, Rene Mantke, Head of Surgery, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: ToPaGe
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Disease
Keywords: Specialization; Pancreatic Surgery; Total Resection; Volume-Outcome-Relationship
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Standard Total pancreatectomy: Total pancreatectomy without vascular or adjacent organ resection. In cases with concomitant liver resection, only an excisional biopsy or wedge resection was to be performed
  Interventions: Procedure: Total pancreatectomy
- Total pancreatectomy with venous resection: Total pancreatectomy with portal vein and/or superior mesenteric vein resection
  Interventions: Procedure: Total pancreatectomy
- Total pancreatectomy with multivisceral resection: Total pancreatectomy with additional adjacent organ resection. The procedure extended beyond pylorus preserving, pylous resecting, and procedures with antrectomy and included the partial or total resection of additional organs with the exception of partial or total splenectomy. Procedures with liver resections, that required a larger atypical, segmental, bisegmental or major (hemihepatectomy) resection.
  Interventions: Procedure: Total pancreatectomy
- Total pancreatectomy with arterial resection: Total pancreatectomy with arterial resection: superior mesenteric artery resections, hepatic artery resections, aortic resections, or resections of the celiac axis
  Interventions: Procedure: Total pancreatectomy

INTERVENTIONS:
Procedure: Total pancreatectomy — Surgical removal of the entire pancreas

SUMMARY:
The purpose of this study was to evaluate the real-world mortality rates of total pancreatectomy across Germany and to understand the impact of hospital caseload on surgical outcomes.

DETAILED DESCRIPTION:
This retrospective observational study analyzed routine data from the nationwide German diagnosis-related group statistics, covering the years 2010 to 2020. The data included all inpatient episodes from acute care hospitals. The study focused on mortality rates associated with total pancreatectomy and examined how these rates varied with the complexity of the surgeries and the volume of procedures performed by different hospitals.

The mortality rates for total pancreatectomy in Germany were found to be more than three times higher than those reported by specialized pancreatic centers. Mortality rates increased significantly with the complexity of the total pancreatectomy procedures, especially those involving arterial resections. Hospitals with lower total pancreatectomy caseloads had higher mortality rates compared to high-volume centers.

Results showed that total pancreatectomies are associated with high mortality rates, particularly in hospitals with lower surgical volumes. The findings suggest that the promising outcomes from specialized centers cannot be generalized to all hospitals performing pancreatic surgeries, highlighting the need for a thorough understanding of the learning curve and specialization in pancreatic surgery to reduce mortality risks.

ELIGIBILITY:
Inclusion Criteria:

* total pancreatectomy between January 2010 and December 2020
* 18 years or older

Exclusion Criteria:

* postmortem pancreatectomy (OPS code 5-525.4)
* removal of a pancreas transplant (OPS code 5-525.3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population encompasses all patients that underwent total pancreatectomy in any German hospital (full survey of the German population).
Sampling Method: Non-Probability Sample
Enrollment: 12938 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Rene Mantke, MD, PhD, Study Director — Head of Surgery at University Hospital Brandenburg an der Havel

IPD SHARING:
Plan to Share IPD: No
No Data is held by the Federal Statistical Office of Germany. Individual participant data is not available for data sharing.